CLINICAL TRIAL: NCT06320535
Title: A Phase 1 Study to Assess the Safety and Immunogenicity of R21/Matrix-M™ Administered in an Escalating Dose, Multi-prime Vaccination Schedule in Healthy Adults
Brief Title: A Phase 1 Study to Assess an Escalating Dose, Multi-prime Vaccination Schedule of R21/Matrix-M™
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC096
Record Dates: First submitted 2024-02-12; First posted 2024-03-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-06

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Intervention Model Description: Participants who opt to receive the escalating dose regimen will be randomized to either Group 1 or Group 2. Recruitment to Groups 1 and 2 will be staggered, as these groups assess a novel administration regimen for R21/Matrix-M:
  * Two participants will be enrolled first, into Group 1 or 2, with a review of safety data collected up to Day 16 by the DSMC.
  * If reactogenicity is acceptable, the remaining participants may be enrolled into Groups 1 and Group 2.
  Participants may be recruited to Group 3 at any time.
  A second DSMC review will take place 16 days after 10 participants have been recruited in Groups 1 and 2 and 5 participants have been recruited in Group 3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Escalating dose R21/Matrix M™ (Experimental): 12 volunteers receiving escalating doses of R21/Matrix M™ adjuvant at days 0, 3, 7, 10, 14, and 56 via intramuscular (IM) injection in the deltoid region of the same arm
  Interventions: Biological: R21/Matrix M™ (Group 1); Procedure: Fine needle aspiration (FNA)
- Group 2: Escalating dose R21/Matrix M™ with delayed booster (Experimental): 12 volunteers receiving escalating doses of R21/Matrix M™ adjuvant at days 0, 3, 7, 10, 14, 168 via intramuscular (IM) injection in the deltoid region of the same arm
  Interventions: Biological: R21/Matrix M™ (Group 2); Procedure: Fine needle aspiration (FNA)
- Group 3: Standard dose R21/Matrix-M™ (Experimental): 12 volunteers receiving two 10mcg doses of R21 in 50mcg of Matrix M™ adjuvant at days 0 and 56 via intramuscular (IM) injection in the deltoid region of the same arm
  Interventions: Biological: R21/Matrix M™ (Group 3); Procedure: Fine needle aspiration (FNA)

INTERVENTIONS:
Biological: R21/Matrix M™ (Group 1) — * 0.50 mcg R21 in 2.75 mcg Matrix-M™ (D0)
  * 0.75 mcg R21 in 3.5 mcg Matrix-M™ (D3)
  * 1.25 mcg R21 in 6.25 mcg Matrix-M™ (D7)
  * 2.5 mcg R21 in 12.5 mcg Matrix-M™ (D10)
  * 5 mcg R21 in 25 mcg Matrix-M™ (D14)
  * 10 mcg R21 in 50 mcg Matrix-M™ (D56)
  Arms: Group 1: Escalating dose R21/Matrix M™
Biological: R21/Matrix M™ (Group 2) — * 0.50 mcg R21 in 2.75 mcg Matrix-M™ (D0)
  * 0.75 mcg R21 in 3.5 mcg Matrix-M™ (D3)
  * 1.25 mcg R21 in 6.25 mcg Matrix-M™ (D7)
  * 2.5 mcg R21 in 12.5 mcg Matrix-M™ (D10)
  * 5 mcg R21 in 25 mcg Matrix-M™ (D14)
  * 10 mcg R21 in 50 mcg Matrix-M™(D168)
  Arms: Group 2: Escalating dose R21/Matrix M™ with delayed booster
Biological: R21/Matrix M™ (Group 3) — * 10 mcg R21 in 50 mcg Matrix-M™ (D0)
  * 10 mcg R21 in 50 mcg Matrix-M™ (D56)
  Arms: Group 3: Standard dose R21/Matrix-M™
Procedure: Fine needle aspiration (FNA) — Participants in all groups will undergo fine needle aspiration (FNA) of axillary lymph nodes draining vaccination site on Day 77 and Day 105 after initial vaccination.

SUMMARY:
This is a phase I clinical study that aims to assess the safety and immunogenicity of a novel, escalating dose regimen of R21/Matrix-M™ in healthy, malaria-naïve adults.

DETAILED DESCRIPTION:
This is a study to assess safety and immunogenicity of a novel dosing regimen for R21/ Matrix-M™, a leading Plasmodium falciparum malaria vaccine, in healthy, malaria-naïve adults. Participants in the study will receive either 6 escalating doses (groups 1 and 2) or 2 standard doses (group 3) of R21/ Matrix-M™, all delivered in the same arm. Up to 36 volunteers will be enrolled and followed up for 12-24 months after their first vaccine.

In addition to blood sampling throughout the follow-up period, participants will undergo fine needle aspiration of axillary lymph nodes twice during the study, to allow further characterisation of immune responses to this novel vaccine regimen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18 to 50 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Participants of childbearing potential only: must practice continuous effective contraception until the last study visit.
* Agreement to refrain from blood donation for the duration of the study.
* Able and willing to provide written informed consent to participate in the trial.

Exclusion Criteria:

* History of clinical malaria (any species) or previous participation in any malaria vaccine trial or controlled human malaria infection trial.
* Travel to a clearly malaria endemic locality during the study period or within the preceding six months, as per the CDC website: https://www.cdc.gov/malaria/travelers/country_table/a.html
* Participation in another research study involving receipt of an investigational medicinal product (IMP) in the 30 days preceding enrolment or 5 half-lives of the investigational medicinal product, whichever is longer, or planned participation during the study period.
* Prior receipt of an IMP likely to impact interpretation of the trial data, as assessed by the Investigator.
* Receipt of any vaccine within 30 days of a study vaccine, with the exception of COVID-19 vaccination.
* Receipt of oral or systemic immunosuppressant medication for more than 14 days in the six months preceding enrolment.
* Receipt of immunoglobulins or blood products (e.g. blood transfusion) in the three months preceding enrolment.
* History of anaphylaxis to vaccination, or allergy likely to be exacerbated by any component of the vaccine or study procedures, including allergy to lidocaine
* Pregnancy, lactation or intention to become pregnant during the study.
* Clinically significant history of chronic disease, including cancer (except basal cell carcinoma or cervical carcinoma in situ), immunodeficiency (including HIV), autoimmune conditions (except mild psoriasis, well-controlled autoimmune thyroid disease, vitiligo or stable coeliac disease), psychiatric disorder, drug or alcohol abuse
* Positive Hepatitis B surface antigen (HBsAg), HIV antibodies or Hepatitis C (HCV) antibodies (except previous HCV vaccine study participants)
* HEMStop score > or = to 2(30) with abnormal coagulation screen or clinical concern regarding bleeding risk.
* Use of medications that increase the risk of bleeding, as assessed by the clinician, including: warfarin, oral antithrombin agents (e.g. Apixaban), low molecular weight heparin
* Any clinically significant abnormality of screening examination, blood or urine tests
* Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may put the volunteer at risk, affect the volunteer's ability to participate in the study or impair interpretation of the study data
* Participants unable to be closely followed for social, geographic or psychological reasons.
* Investigator inability to corroborate a participant's medical history via access to NHS electronic records and/or their GP.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety of R21/Matrix-M™ administered in an escalating dose, multi prime vaccination schedule versus a standard prime-boost regimen in healthy UK adults, measured by the number of solicited adverse events in each group | 7 days post-vaccination
  Occurrence of solicited local and systemic reactogenicity signs and symptoms will be collected for 7 days following each vaccination. Solicited adverse event data will be tabulated, detailing frequency, duration and severity of the AEs.
Safety of R21/Matrix-M™ administered in an escalating dose, multi prime vaccination schedule versus a standard prime-boost regimen in healthy UK adults, measured by the number of unsolicited adverse events and laboratory adverse events in each group | 28 days post-vaccination.
  Occurrence of unsolicited adverse events and changes from baseline in laboratory safety measures will be collected for 28 days following each vaccination. Unsolicited AE data will be tabulated, detailing frequency, duration and severity of AEs. Hematological and biochemical laboratory values will be presented according to local grading scales.
Safety of R21/Matrix-M™ administered in an escalating dose, multi prime vaccination schedule versus a standard prime-boost regimen in healthy UK adults, measured by the number of serious adverse events in each group | For the follow-up period of the study, between 1-2 years
  Occurrence of serious adverse events (SAEs), adverse events of special interest (AESIs) and withdrawal due to AE(s)/SAE(s) will be described in detail.
Humoral immunogenicity of R21/Matrix-M™ administered in an escalating dose, multi-prime vaccination schedule verus a standard prime-boost regimen in healthy UK adults | For the follow-up period of the study, between 1-2 years
  Antibody dynamics will be assessed by measuring NANP-IgG at baseline and various timepoints during the trial.

OTHER OUTCOMES:
Impact of vaccination schedule on immune response in participants vaccinated with R21/Matrix-M™ administered in escalating dose, multi-prime vaccination schedules versus a standard prime-boost regimen | For the follow-up period of the study, between 1-2 years
  (Exploratory outcome measure) Exploratory immunology to further investigate the relationship between cellular and humoral immunity and vaccine regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Hodgson, DPhil FRCP, Principal Investigator — Center for Clinical Vaccinology and Tropical Medicine, University of Oxford; Rajeka Lazarus, DPhil FRCP, Principal Investigator — University Hospitals Bristol and Weston Foundation Trust
Locations (2):
- United Kingdom (2):
  - Centre for Clinical Vaccinology and Tropical Meducine, Churchill Hospital, University of Oxford, Oxford, Oxfordshire
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol